CLINICAL TRIAL: NCT05785806
Title: Construction and Effect Evaluation of Parent Infant Skin-to-Skin Contact Intervention Program Based on The Co-parenting Theory
Brief Title: Parent Infant Skin-to-Skin Contact Intervention Based on The Co-parenting Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, chen xiao, Chief Physician of Anesthesiology, Affiliated Hospital of Jiangnan University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JNU20221201IRB20
Record Dates: First submitted 2023-03-02; First posted 2023-03-27 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Anxiety; Parturition; Precipitate
Keywords: Paternity; Skin-to-skin contact; Co-parenting; Parents' psychological health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Skin to skin contact and co-parenting theory course (Experimental): 1. Skin to skin contact and co-parenting theory course
  2. Skin to skin contact instruction manual and co-parenting theory brochure
  3. Daily face-to-face skin to skin contact guidance during hospitalization
  4. Online punching skin to skin contact
  Interventions: Behavioral: Skin to skin contact and co-parenting theory course; Behavioral: Skin to skin contact instruction manual and co-parenting theory brochure; Behavioral: Daily face-to-face skin to skin contact guidance during hospitalization; Behavioral: Online punching skin to skin contact
- Routine obstetric care (Other): Routine prenatal training and postpartum education, including basic breastfeeding guidelines, touching, etc.
  Interventions: Behavioral: Routine obstetric care

INTERVENTIONS:
Behavioral: Skin to skin contact and co-parenting theory course — On the day before delivery, pregnant women and their husbands attend a course on the theory of skin contact and co-parenting to explain the role and importance of skin contact ; to understand the knowledge of co-parenting and parenting care ; to learn the communication method and future parenting plan based on the theory of co-parenting, and to learn the operation of skin contact with newborns after delivery.
  Arms: Skin to skin contact and co-parenting theory course
Behavioral: Skin to skin contact instruction manual and co-parenting theory brochure — According to reading and analyzing the literature on skin contact, summarize the content of skin contact operation guidance ; read and analyze the relevant literature of co-parenting theory, and summarize the theoretical knowledge and practical operation methods of co-parenting. Pregnant women and their spouses can check in time.
  Arms: Skin to skin contact and co-parenting theory course
Behavioral: Daily face-to-face skin to skin contact guidance during hospitalization — After delivery, face-to-face skin-to-skin contact guidance and co-parenting communication and practice were given to the parturient and her husband on a daily basis during hospitalization. Establish a daily fixed skin contact duration target, and the specific operation is freely allocated by both parents.
  Arms: Skin to skin contact and co-parenting theory course
Behavioral: Online punching skin to skin contact — Share common parenting related knowledge, daily skin contact reminders, emphasize mutual recognition and mutual support of parents, and conduct WeChat follow-up every two weeks to understand the physical and mental status of both parties and the growth of infants.
  Arms: Skin to skin contact and co-parenting theory course
Behavioral: Routine obstetric care — Routine prenatal training and postpartum education, including basic breastfeeding guidelines, touching, etc.
  Arms: Routine obstetric care

SUMMARY:
The goal of this clinical intervention study is to construct a neonatal skin contact program for cesarean section primipara families with the cooperation of both parents.So as to provide theoretical basis and practical guidance for pregnant women and their spouses, and reduce the possibility of anxiety and depression of pregnant women and their spouses. Promoting the ability of fathers to participate in co-parenting can help mothers and their spouses adapt to the new role of ' parents ' and enhance their sense of parenting competence and happiness. The main questions it aims to answer are:

* How to publicize and educate knowledge about co-parenting theory and skin contact knowledge and use the co-parenting theory to design a suitable skin contact scheme?
* What are the benefits of skin to skin contact between parents after cesarean section?

  1. Participants will take prenatal classes on co-parenting and skin to skin contact.
  2. Participants will receive brochures on co-parenting theory and skin to skin contact.
  3. Participants will receive face-to-face skin-to-skin contact guidance every day during postpartum hospitalization to correctly perform skin to skin contact.
  4. Participants will be online to punch in skin contact. There is a comparison group: routine prenatal and post-natal care without additional educational support.

Researchers will compare the comparison group to see the cesarean section parents in the postpartum distribution of skin contact tasks, joint skin contact, whether will the intimate relationship between parents and infants, parents ' mental health, anxiety level.

DETAILED DESCRIPTION:
Through pre-clinical research, it was found that primipara families lacked guidance and intervention for fathers, and theoretical basis and practical guidance were needed to build a new family system at the first time after delivery. Pregnant women need the support and help of their spouses or family members in the critical period of physical and mental recovery after delivery ; the newborn needs daily life care, interactive communication and caring companionship to meet the physical, emotional and psychological needs of the baby ; the parental participation of primipara spouses is at a low level. Maternal spouses lack relevant knowledge and experience, and need targeted guidance and intervention to promote their parental participation.

After the mother underwent cesarean section, due to physical factors such as pain and fetal crying, the mother 's mood is affected, and the arrival of a new life is full of anxiety, which will lead to problems in the mother 's lactation. Production and childrearing are not the task of the mother alone. The purpose of this study is to let the father participate in childrearing at the first time after childbirth, and what are the benefits to the family.

ELIGIBILITY:
Inclusion Criteria:

* Primipara
* cesarean section
* 37-42 weeks of pregnancy
* junior high school education or above
* Couples live together
* Both husband and wife can recognize and understand Chinese

Exclusion Criteria:

* multiple pregnancy
* Pregnant women have serious complications / complications, such as eclampsia, postpartum hemorrhage, severe cardiopulmonary dysfunction, etc.
* Prenatal examination of the fetus with chromosomal abnormalities or possible malformations
* One of the couple has mental retardation or mental disorders can not cooperate
* Delivery before 37 weeks of gestation
* Postpartum mother-to-child separation, newborns need to be treated and monitored in NICU
* Evaluation information collection is not perfect

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 111 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-10-21 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Postpartum parents ' sense of security (Postpartum Parental Safety Scale，PPSS) | one week after delivery
  Postpartum Parental Safety Scale，PPSS is a survey tool used to assess the sense of security of both parents after childbirth, and to assess the sense of security of parents in the first week after delivery.The Chinese version of PPSS scale is divided into mother version and father version.The PPSS mother version had 18 items and the father version had 13 items, all of which were scored using a four-level scoring method ( 1-4 points ). Mother version of the scale minimum score of eighteen points, the highest score of seventy-two ; the minimum score of the father 's version scale is 13 points, and the maximum score is 52 points.The answer options ranged from ' very disagree ' to ' very agree '. The higher the score, the higher the sense of security.
Co-parenting situation (The Brief Coparenting Relationship Scale， Brief CRS ) | 42 days and three months after delivery
  The Brief Coparenting Relationship Scale ( Brief CRS ) was jointly developed by Feinberg, Brown and Kan in 2012. The scale uses a self-reported approach to comprehensively assess the quality of coparenting in a family. It consists of 14 items and 7 subscales.The Brief Coparenting Relationship Scale can be used as a tool to measure the effect of father in coparenting in Chinese family． The scale can be used to measure father's support and involvement with breastfeeding in the study of breastfeeding．All items were scored by Likert 7, of which 3 items were reverse scoring, with a total score of 0-84. The higher the score, the better the co-parenting, that is, the stronger the father 's support.
Maternal and infant attachment | 42 days and three months after delivery
  The Maternal Postnatal Attachment Scale ( MPAS ) is a self-reported scale developed by Condon and Corkindale to reflect the degree of subjective emotional connection between mothers and their infants.The Maternal Postnatal Attachment Scale is a valid and reliable tool for the evaluation of the early affectionate mother-infant relationship.The scale has 18 items, including two, three, four and five options.The total score span of the scale is between 18-90, and the higher the score, the higher the level of maternal and child attachment.
Father-infant attachment | 42 days and three months after delivery
  Father-infant attachment will be evaluated by the use of the Paternal Postnatal Attachment Scale (PPAS) originally designed by John T. Condon and colleagues. This is a 19-item, self-report questionnaire including three subscales: patience and tolerance, pleasure in interaction, and affection and pride.The total score span of the scale is between 19-95, and the higher the score, the higher the level of attachment between father and baby.
Neonatal Behaviral Neurological Assessment，NBNA | 3 days and 42 days after delivery
  French Ameil Tison neonatal neuromotor examination method, combined with the specific situation in China.It is also of great significance for understanding the behavioral abilities of newborns, promoting early development of eugenics and intellectual cognition.NBNA examination is divided into five parts, including six items of neonatal behavioral ability, four items of passive muscle tone, four items of active muscle tone, three items of Primitive reflexes, and three items of general response, with a total of 40 points. The higher the score, the better the behavioral neurological function.

SECONDARY OUTCOMES:
The anxiety level | one week,42 days and three months after delivery
  The Self-Rating Anxiety Scale,SAS will be used by both parents to assess the anxiety levels.The self-rating anxiety scale compiled by Zung in 1971 is a self-rating scale, which is used to evaluate the subjective feelings of adults and the degree of anxiety. The scale includes 20 items, including 15 positive scores and 5 negative scores. According to the frequency of symptoms defined by the item, the Likert 4-level scoring method was used. From ' no or little time ' to ' most or all of the time ', the positive scoring questions were rated as 1-4 points, and the reverse scoring questions were rated as 4-1 points. Standard score = total coarse score * 1.25, take the integer part, with SAS standard as the cut-off value, the cut-off value is less than 50 points for no anxiety group, 50 ~ 59 points for mild anxiety group, 60 ~ 69 points for moderate anxiety group, 69 points or more for severe anxiety group.
The depression level | one week,42 days and three months after delivery
  The Self-Rating Depression Scale,SDS will be used by both parents to assess the depression level.Self-Rating Depression Scale ( SDS ) is a self-rating scale compiled by Zung in 1965, which is used to evaluate the subjective feelings of adults and the severity of depression. It includes 20 items, using a 4-level score, 10 positive score items, and 10 reverse score items. The total rough score was obtained by adding the scores of 20 items. The standard score = total rough score * 1.25, and the integer part was taken. The standard value of SDS was divided into the boundary value. The boundary value was less than 53, which was divided into the non-depression group, 53-62 was divided into the mild depression group, 63-72 was divided into the moderate depression group, and more than 72 was the severe depression group.

CONTACTS AND LOCATIONS:
Overall Officials: Xuejun Tian, Study Director — Head Nurse of Obstetrics at Jiangnan University Affiliated Hospital; Lingxia Kong, Study Chair — A student of Wuxi Medical College Jiangnan University; Xiao Chen, Doctor, Study Director — Professor at Jiangnan University; Yuting Jiang, Principal Investigator — A student of Wuxi Medical College Jiangnan University; Chunting Li, Study Chair — A student of Wuxi Medical College Jiangnan University; Qian Wang, Study Chair — A student of Wuxi Medical College Jiangnan University; Xian Ding, Doctor, Study Director — Associate Professor at Jiangnan University
Locations (1):
- Medical College Jiangnan University, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feinberg ME, Brown LD, Kan ML. A Multi-Domain Self-Report Measure of Coparenting. Parent Sci Pract. 2012 Jan 1;12(1):1-21. doi: 10.1080/15295192.2012.638870. Epub 2012 Jan 20. PMID 23166477
- [Background] Schoppe-Sullivan SJ, Weldon AH, Cook JC, Davis EF, Buckley CK. Coparenting behavior moderates longitudinal relations between effortful control and preschool children's externalizing behavior. J Child Psychol Psychiatry. 2009 Jun;50(6):698-706. doi: 10.1111/j.1469-7610.2008.02009.x. Epub 2009 Jan 21. PMID 19207627
- [Background] Takeishi Y, Nakamura Y, Kawajiri M, Atogami F, Yoshizawa T. Developing a Prenatal Couple Education Program Focusing on Coparenting for Japanese Couples: A Quasi-Experimental Study. Tohoku J Exp Med. 2019 Sep;249(1):9-17. doi: 10.1620/tjem.249.9. PMID 31511452
- [Background] Woody CA, Ferrari AJ, Siskind DJ, Whiteford HA, Harris MG. A systematic review and meta-regression of the prevalence and incidence of perinatal depression. J Affect Disord. 2017 Sep;219:86-92. doi: 10.1016/j.jad.2017.05.003. Epub 2017 May 8. PMID 28531848
- [Background] Cameron EE, Sedov ID, Tomfohr-Madsen LM. Prevalence of paternal depression in pregnancy and the postpartum: An updated meta-analysis. J Affect Disord. 2016 Dec;206:189-203. doi: 10.1016/j.jad.2016.07.044. Epub 2016 Jul 20. PMID 27475890
- [Background] Philpott LF, Corcoran P. Paternal postnatal depression in Ireland: Prevalence and associated factors. Midwifery. 2018 Jan;56:121-127. doi: 10.1016/j.midw.2017.10.009. Epub 2017 Oct 20. PMID 29096280
- [Background] Moneta C ME. [Attachment and loss: rediscovering John Bowlby]. Rev Chil Pediatr. 2014 Jun;85(3):265-8. doi: 10.4067/S0370-41062014000300001. No abstract available. Spanish. PMID 25697242
- [Background] Kerns KA, Brumariu LE. Is Insecure Parent-Child Attachment a Risk Factor for the Development of Anxiety in Childhood or Adolescence? Child Dev Perspect. 2014 Mar 1;8(1):12-17. doi: 10.1111/cdep.12054. PMID 24660023
- [Background] Benoit D. Infant-parent attachment: Definition, types, antecedents, measurement and outcome. Paediatr Child Health. 2004 Oct;9(8):541-545. doi: 10.1093/pch/9.8.541. PMID 19680481
- [Background] Feinberg ME, Kan ML. Establishing family foundations: intervention effects on coparenting, parent/infant well-being, and parent-child relations. J Fam Psychol. 2008 Apr;22(2):253-63. doi: 10.1037/0893-3200.22.2.253. PMID 18410212
- [Background] Feinberg ME, Jones DE, Hostetler ML, Roettger ME, Paul IM, Ehrenthal DB. Couple-Focused Prevention at the Transition to Parenthood, a Randomized Trial: Effects on Coparenting, Parenting, Family Violence, and Parent and Child Adjustment. Prev Sci. 2016 Aug;17(6):751-64. doi: 10.1007/s11121-016-0674-z. PMID 27334116
- [Background] Izett E, Rooney R, Prescott SL, De Palma M, McDevitt M. Prevention of Mental Health Difficulties for Children Aged 0-3 Years: A Review. Front Psychol. 2021 Sep 29;11:500361. doi: 10.3389/fpsyg.2020.500361. eCollection 2020. PMID 34777074
- [Background] Allport-Altillo BS, Aqil AR, Nelson T, Johnson SB, Labrique AB, Carabas Y, Marcell AV. Parents' Perspectives on Supporting Father Involvement in African American Families During Pregnancy and Early Infancy. J Natl Med Assoc. 2020 Aug;112(4):344-361. doi: 10.1016/j.jnma.2020.04.002. Epub 2020 May 11. PMID 32409095
- [Background] Shorey S, Dennis CL, Bridge S, Chong YS, Holroyd E, He HG. First-time fathers' postnatal experiences and support needs: A descriptive qualitative study. J Adv Nurs. 2017 Dec;73(12):2987-2996. doi: 10.1111/jan.13349. Epub 2017 Jun 21. PMID 28557020
- [Background] Shorey S, Lau Y, Dennis CL, Chan YS, Tam WWS, Chan YH. A randomized-controlled trial to examine the effectiveness of the 'Home-but not Alone' mobile-health application educational programme on parental outcomes. J Adv Nurs. 2017 Sep;73(9):2103-2117. doi: 10.1111/jan.13293. Epub 2017 Apr 7. PMID 28276086
- [Background] Jarjour IT. Neurodevelopmental outcome after extreme prematurity: a review of the literature. Pediatr Neurol. 2015 Feb;52(2):143-52. doi: 10.1016/j.pediatrneurol.2014.10.027. Epub 2014 Nov 4. PMID 25497122
- [Background] Baron IS, Litman FR, Ahronovich MD, Baker R. Late preterm birth: a review of medical and neuropsychological childhood outcomes. Neuropsychol Rev. 2012 Dec;22(4):438-50. doi: 10.1007/s11065-012-9210-5. Epub 2012 Aug 7. PMID 22869055
- [Background] Mori R, Khanna R, Pledge D, Nakayama T. Meta-analysis of physiological effects of skin-to-skin contact for newborns and mothers. Pediatr Int. 2010 Apr;52(2):161-70. doi: 10.1111/j.1442-200X.2009.02909.x. Epub 2009 Jun 11. PMID 19519670
- [Background] Feldman R, Eidelman AI. Skin-to-skin contact (Kangaroo Care) accelerates autonomic and neurobehavioural maturation in preterm infants. Dev Med Child Neurol. 2003 Apr;45(4):274-81. doi: 10.1017/s0012162203000525. PMID 12647930
- [Background] Ferber SG, Makhoul IR. The effect of skin-to-skin contact (kangaroo care) shortly after birth on the neurobehavioral responses of the term newborn: a randomized, controlled trial. Pediatrics. 2004 Apr;113(4):858-65. doi: 10.1542/peds.113.4.858. PMID 15060238
- [Background] Charpak N, Ruiz JG, Zupan J, Cattaneo A, Figueroa Z, Tessier R, Cristo M, Anderson G, Ludington S, Mendoza S, Mokhachane M, Worku B. Kangaroo Mother Care: 25 years after. Acta Paediatr. 2005 May;94(5):514-22. doi: 10.1111/j.1651-2227.2005.tb01930.x. PMID 16188735
- [Background] Pillai Riddell RR, Racine NM, Gennis HG, Turcotte K, Uman LS, Horton RE, Ahola Kohut S, Hillgrove Stuart J, Stevens B, Lisi DM. Non-pharmacological management of infant and young child procedural pain. Cochrane Database Syst Rev. 2015 Dec 2;2015(12):CD006275. doi: 10.1002/14651858.CD006275.pub3. PMID 26630545
- [Background] Feldman R, Eidelman AI, Sirota L, Weller A. Comparison of skin-to-skin (kangaroo) and traditional care: parenting outcomes and preterm infant development. Pediatrics. 2002 Jul;110(1 Pt 1):16-26. doi: 10.1542/peds.110.1.16. PMID 12093942
- [Background] Anderzen-Carlsson A, Lamy ZC, Eriksson M. Parental experiences of providing skin-to-skin care to their newborn infant--part 1: a qualitative systematic review. Int J Qual Stud Health Well-being. 2014 Oct 13;9:24906. doi: 10.3402/qhw.v9.24906. eCollection 2014. PMID 25319746
- [Background] Velandia M, Uvnas-Moberg K, Nissen E. Sex differences in newborn interaction with mother or father during skin-to-skin contact after Caesarean section. Acta Paediatr. 2012 Apr;101(4):360-7. doi: 10.1111/j.1651-2227.2011.02523.x. Epub 2011 Dec 1. PMID 22077187
- [Background] Erlandsson K, Dsilna A, Fagerberg I, Christensson K. Skin-to-skin care with the father after cesarean birth and its effect on newborn crying and prefeeding behavior. Birth. 2007 Jun;34(2):105-14. doi: 10.1111/j.1523-536X.2007.00162.x. PMID 17542814
- [Background] Shorey S, He HG, Morelius E. Skin-to-skin contact by fathers and the impact on infant and paternal outcomes: an integrative review. Midwifery. 2016 Sep;40:207-17. doi: 10.1016/j.midw.2016.07.007. Epub 2016 Jul 5. PMID 27476026
- [Background] Erlandsson K, Christensson K, Fagerberg I. Fathers' lived experiences of getting to know their baby while acting as primary caregivers immediately following birth. J Perinat Educ. 2008 Spring;17(2):28-36. doi: 10.1624/105812408X298363. PMID 19252686
- [Background] Makela H, Axelin A, Feeley N, Niela-Vilen H. Clinging to closeness: The parental view on developing a close bond with their infants in a NICU. Midwifery. 2018 Jul;62:183-188. doi: 10.1016/j.midw.2018.04.003. Epub 2018 Apr 11. PMID 29684798
- [Background] Olsson E, Eriksson M, Anderzen-Carlsson A. Skin-to-Skin Contact Facilitates More Equal Parenthood - A Qualitative Study From Fathers' Perspective. J Pediatr Nurs. 2017 May-Jun;34:e2-e9. doi: 10.1016/j.pedn.2017.03.004. Epub 2017 Mar 29. PMID 28364962
- See also: A website providing emotional guidance and support for new parents — http://www.panda.org.au/info-support/after-birth/contributingfactors-for-postnatal-depression-or-anxiety

DOCUMENTS (1):
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT05785806/ICF_001.pdf